CLINICAL TRIAL: NCT00822276
Title: Pilot Study To Determine The Underlying Mechanisms For Infection And Colonization By Staphylococcus Aureus Of The Skin Of Atopic Dermatitis Subjects With And Without A History Of Eczema Herpeticum (ADVN MRSA 10)
Brief Title: The Underlying Mechanisms For S. Aureus Infection And Colonization Of Skin in People With Atopic Dermatitis With And Without Eczema Herpeticum (MRSA)
Acronym: MRSA
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ADVN MRSA 10
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus; Atopic Dermatitis; Eczema Herpeticum; MRSA
Keywords: Methicillin-resistant Staphylococcus aureus; MRSA; Methicillin-sensitive Staphylococcus aureus; MSSA; Atopic Dermatitis; Eczema Herpeticum
MeSH Terms: conditions — Dermatitis, Atopic; Kaposi Varicelliform Eruption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs, skin swabs, tape strippings, and blood draws.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- ADEH+ participants colonized with MSSA
- ADEH+ participants colonized with MRSA
- Uncolonized ADEH+ participants
- ADEH- participants colonized with MSSA
- ADEH- participants colonized with MRSA
- Uncolonized ADEH- subjects
- Non-atopic uncolonized S. aureus participants

SUMMARY:
Staphylococcus aureus (S.aureus) is a bacterium that causes many painful skin and soft tissue conditions, such as scalded-skin syndrome, boils, or impetigo. Serious cases may result in deadly complications but S.aureus can usually be treated successfully with antibiotics. There are, however, certain strains which cannot be treated with standard antibiotics. Methicillin-resistant staphylococcus aureus (MRSA) is one such strain.

MRSA is increasingly being seen in both hospital and community settings, making it a serious public health issue. People with Atopic Dermatitis (AD), particularly those with a history of Eczema Herpeticum (EH), may be at greater risk for infection by MRSA. The reason for this higher risk is unknown but may be linked to extended treatment with staphylococcus antibiotics in addition to the absence of certain proteins on their skin, which have immune function. The purpose of this study is to determine the reasons for MRSA infection in AD participants with and without a history of EH.

DETAILED DESCRIPTION:
The emergence of drug-resistant staphylococcal strains was first seen in the US almost a decade ago, when the Centers for Disease Control (CDC) reported four fatal community-based MRSA infections in children. In recent years, MRSA has grown into a serious public health concern with an increasing number of both hospital-acquired and community-acquired cases being seen.

There will be approximately 130 participants recruited for this trial. The study population will consist of people with Atopic Dermatitis (AD) and people without Atopic Dermatitis (non-atopic). AD is a skin disorder with an itchy, red skin rash. People with AD are more likely to get bacterial and viral skin infections, possibly because they lack certain proteins in their skin, which help the body's immune system to fight infections. AD people with a history of Eczema Herpeticum (EH) may also be at greater risk for being infected with MRSA. This could be due to extended treatment courses with staphylococcal antibiotics, especially because overuse and misuse of antibiotics can lead to bacterial antibiotic resistance. The precise reasons are unknown. The purpose of this study is to determine the reasons for infection in AD participants with and without a history of EH.

Investigators are seeking to recruit patients with either Methicillin-sensitive staphylococcus aureus (MSSA) or MRSA bacteria on their skin, so that they may adequately study potential factors related to MRSA infection.

Investigators will determine if the MRSA collected from people with AD is primarily community or hospital associated. They will also determine if the proteins on the skin of ADEH+ people with MRSA differ from the proteins on the skin of AD people with MSSA or people without AD, or if there are any marked differences in serum total IgE levels between AD subjects with MRSA, MSSA, or without S. aureus. Approximately 60 ADEH+ and 60 ADEH- participants will need to be enrolled to find participants with MRSA or MSSA on their skin. Presence of these bacteria on the skin can only be determined once skin swabs are collected and tested.

If participants are deemed eligible at screening, they will continue on to the study visit, which will last for approximately 2-3 hours. At the study visit, participants will be asked to provide information related to their medical history including infection, hospitalization, and medication record. Additionally, a skin exam will be performed to verify diagnosis (ADEH-, ADEH+, or non-atopic); nasal and skin swabs samples will be collected; tape strippings samples will be collected; and a blood sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Parent, or legal guardian willing to provide informed consent, if necessary
* Residing in the U.S.
* Have active AD with or without a history of EH as diagnosed using the ADVN Standardized Diagnostic Criteria OR are non-atopic as diagnosed using the ADVN Standardized Diagnostic Criteria

Exclusion Criteria:

* History of any systemic illness (i.e., immunodeficiency disorders such as human immunodeficiency virus [HIV] or lupus erythematosus) other than the condition being studied
* Presence of active systemic malignancy, excluding uncomplicated non-melanoma skin cancer
* Presence of any skin disease other than AD that might compromise the stratum corneum barrier (e.g., bullous disease, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome])
* Use of topical medications including (but not limited to) Elidel, Protopic, or topical corticosteroids at the site of the skin lesion within the last 3 days
* Use of topical antibiotics within the last 24 hours
* Use of oral antibiotics within the last 10 days. Subjects who are known to be culture positive for MSSA or MRSA despite antibiotic treatment will not be excluded.
* History of serious or life-threatening reactions to tape or adhesives will be excluded from the tape stripping procedure

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ADEH-, ADEH+ people who may or may not be colonized with MRSA or MSSA, and non-atopic people not colonized with MRSA or MSSA.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
MRSA isolates from nasal and/or skin swabs will be characterized as either nosocomial or community-associated | At Study Entry

SECONDARY OUTCOMES:
Proteomic profiling will be conducted on taped stripped skin samples of lesional and non-lesional skin in order to identify potential biomarkers associated with susceptibility to MRSA colonization. Metabolomic profiling may be conducted pending funding. | At Study Entry
Genomic analyses of superficial bacterial flora from lesional and non-lesional skin swab samples | At Study Entry

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD, PhD, Principal Investigator — National Jewish Health; Richard Gallo, MD, PhD, Principal Investigator — University of California, San Diego; Gloria David, PhD, MHSc, Principal Investigator — Rho, Inc.; Patrick Schlievert, PhD, Principal Investigator — University of Minnesota; Nichole Reisdorph, PhD, MS, Principal Investigator — National Jewish Health
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado

REFERENCES:
- [Result] Schlievert PM, Case LC, Strandberg KL, Abrams BB, Leung DY. Superantigen profile of Staphylococcus aureus isolates from patients with steroid-resistant atopic dermatitis. Clin Infect Dis. 2008 May 15;46(10):1562-7. doi: 10.1086/586746. PMID 18419342
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/